CLINICAL TRIAL: NCT04883996
Title: A Phase 1/2, Randomized, Placebo Controlled Crossover Study to Assess the Safety, Pharmacodynamics, and Efficacy of EXP039 Ophthalmic Solution in Participants With Myopia or Hyperopia
Brief Title: A Phase 1/2 Crossover Study to Assess EXP039 for Myopia or Hyperopia
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Canyon City Eyecare (Other)
Collaborators: Nevakar, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CP-EXP039-0001
Record Dates: First submitted 2021-05-07; First posted 2021-05-12 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-05

CONDITIONS: Hyperopia; Myopia
Keywords: Hyperopia; Myopia; Visual Acuity; Mesopic
MeSH Terms: conditions — Hyperopia; Myopia | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- EXP039 (Active Comparator): At Visit 1, single dose 1 drop of EXP039 1% is adminstered, followed by washout period of 1-10 days. Subsequently, subjects will crossover to single dose 1 drop saline at Visit 2.
  Interventions: Drug: 1% EXP039
- Saline control (Placebo Comparator): At Visit 1, single dose 1 drop of saline is adminstered, followed by washout period of 1-10 days. Subsequently, subjects will crossover to single dose 1 drop EXP039 1% at Visit 2.
  Interventions: Other: Saline control

INTERVENTIONS:
Drug: 1% EXP039 — 1% EXP039 (commercially available as Isopto® Carpine) contains 1% active ingredient (10 mg/mL),
  Other Names: Isopto® Carpine
  Arms: EXP039
Other: Saline control — Saline
  Other Names: Saline
  Arms: Saline control

SUMMARY:
Assess the Safety, Pharmacodynamics, and Efficacy of EXP039 Ophthalmic Solution in Participants with Myopia or Hyperopia

DETAILED DESCRIPTION:
To characterize the effect of pupillary miosis as achieved with EXP039 1% ophthalmic solution in terms of mean number of lines (Early Treatment Diabetic Retinopathy Study [ETDRS]) of improvement from baseline in binocular (both eyes open) mesopic high-contrast uncorrected distance visual acuity (UDVA) at 1-hour post treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 to ≤80 years
2. Participants must be in good general health, with no significant medical problems that, in the opinion of the investigator, would preclude participation in the trial, at Screening and/or before administration of the dose of study drug
3. Low-to-moderate hyperopia (SER of +0.50D to +2.00D) or myopia (SER of -0.50 D to -4.00D) at Screening
4. Between-eye SER difference of no more than 0.50D
5. Best-corrected distance visual acuity better than or equal to 20/20 in both eyes at Screening
6. Astigmatism in each eye of less than or equal to 0.75D with manifest refraction at Screening
7. Women of childbearing potential (WOCBP) must have a negative urine pregnancy test at Screening
8. WOCBP must be non-pregnant and non-lactating, and must use a medically approved, highly effective contraception method from Screening until study completion, including the follow up period. Female participants who are in same sex relationships are not required to use contraception.Males must be surgically sterile (>30 days since vasectomy with no viable sperm), abstinent, or if engaged in sexual relations with a WOCBP, the participant and his partner must use a medically approved, highly effective contraceptive method from Screening until study completion, including the follow-up period.
9. Males must not donate sperm for at least 90 days after the last dose of study drug
10. Participants must have the ability and willingness to attend the necessary visits
11. Participants must be willing and able to provide written informed consent after the nature of the study has been explained and prior to the commencement of any study procedures.

Exclusion Criteria:

1. Any central corneal abnormality (e.g., keratoconus, Pellucid marginal degeneration, corneal scar, Fuchs' endothelial dystrophy, guttata, or edema) in either eye that is likely to interfere with visual acuity
2. Moderate or severe dry eye as defined by corneal fluorescein staining score of ≥3 on Oxford scale at Screening
3. Any clinically significant pupillary or iris abnormality (e.g., anisocoria of >1 mm between eyes at Screening or baseline, abnormal pupil shape in either eye, iris transillumination defects, or any congenital or traumatic defect of the iris)
4. Narrow iridocorneal angles (Shaffer grade ≤2 or lower on gonioscopy examination), history of angle-closure glaucoma, or previous iridotomy
5. Intraocular pressure (IOP) <8 mmHg or >23 mmHg in either eye or history of glaucoma or ocular hypertension
6. Any clinically significant abnormal lens finding (e.g., cataract, loose zonules, exfoliation, pseudoexfoliation)
7. History of any intraocular surgery including cataract surgery or phakic intraocular lens surgery
8. History in either eye of previous corneal inlay, full- or partial-thickness corneal transplant, radial keratotomy or any corneal surgery including laser-based corneal refractive surgery
9. Any clinically significant abnormal finding on dilated fundus examination in either eye or known history of retinal detachment, retinal trauma, retinal or vitreal surgery, or clinically significant retinal disease in either eye
10. Clinically significant strabismus or diplopia
11. History of stereo vision difficulties
12. History of optic neuropathy or amblyopia in either eye
13. Use of orthokeratology contact lenses within the past 1 month prior to EXP039 dosing on Day 1
14. Use of temporary or permanent punctal plugs or history of punctal cautery in one or both eyes
15. Planned use of any contact lenses during the study
16. Allergy to pilocarpine or any of its excipients
17. Serious systemic illness that, in the opinion of the Investigator's, would render the participant ineligible
18. Pre-planned hospitalization or ocular or systemic surgery during the study period
19. History of any substance abuse (alcohol and/or illegal drugs) and not willing to abstain from drug(s) and reasonably limit alcohol consumption to approximately 2 alcoholic beverages per day during the 30-day study period
20. Participation in any other study of investigational therapy during the study period or within the last 30 days or 5 half-lives, whichever is longer
21. Unwilling or unable to complete study procedures or to be followed up for the duration of the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-08-30 (Estimated)

PRIMARY OUTCOMES:
UDVA | 1 hour
  Mesopic high-contrast uncorrected distance visual acuity

CONTACTS AND LOCATIONS:
Overall Officials: Milton Hom, OD FAAO, Principal Investigator — Canyon City Eyecare
Locations (1):
- Canyon City Eyecare, Azusa, California, United States

IPD SHARING:
Plan to Share IPD: No